CLINICAL TRIAL: NCT07349719
Title: Impact of Dynamic Compliance-guided Ventilation on Postoperative Pulmonary Function in Lumbar Stabilization Surgery:A Prospective Study
Brief Title: Dynamic Compliance-Guided Ventilation in Lumbar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Burak NALBANT, Assistant Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1-25-1645
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Spine Stenosis; Lumbar Disc Herniation; Ventilator-Induced Lung Injury; Postoperative Complications
MeSH Terms: conditions — Intervertebral Disc Displacement; Ventilator-Induced Lung Injury; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Compliance Guided Ventilation (Active Comparator): Patients receive intraoperative ventilation adjusted according to real time dynamic compliance monitoring
  Interventions: Procedure: Dynamic Compliance Guided Ventilation
- Standart Ventilation (Active Comparator): Patients receive intraoperative ventilation based on conventional standart settings without dynamic compliance adjustment
  Interventions: Procedure: Standard Ventilation

INTERVENTIONS:
Procedure: Dynamic Compliance Guided Ventilation — After intubation and prone positioning, both groups will undergo the same initial recruitment maneuver as described above. In the dynamic compliance-guided group, positive end expiratory pressure(PEEP) will then be titrated according to dynamic compliance (Cdyn = VT / [Ppeak - PEEP])(Ppeak: Peak airway pressure)(VT:Tidal volume). Tidal volume will be set at 7 ml/kg, respiratory rate 12/min, and positive end expiratory pressure(PEEP) reduced stepwise from 20 cmH₂O to 5 cmH₂O in increments of 2 cmH₂O. Each positive end expiratory pressure(PEEP) level (19, 17, 15, 13, 11, 9, 7, 5 cmH₂O) will be maintained for 10 respiratory cycles, with Cdyn measured at the end of each level. The positive end expiratory pressure(PEEP) corresponding to the highest dynamic compliance will be selected and maintained throughout the surgery.In both groups, a 30% t-pause will be applied throughout the operation after intubation. Patients will be ventilated in volume-controlled ventilation (VCV) mode.
  Arms: Dynamic Compliance Guided Ventilation
Procedure: Standard Ventilation — After intubation, both groups will initially receive conventional ventilation in volume-controlled mode with a tidal volume of 7 ml/kg (predicted body weight), positive end expiratory pressure(PEEP) of 5 cmH₂O, and an inspiratory-to-expiratory ratio of 1:2. Respiratory rate will be adjusted to maintain end-tidal CO₂ between 35-45 mmHg. Following prone positioning, a recruitment maneuver will be performed using pressure-controlled ventilation, gradually increasing positive end expiratory pressure(PEEP) from 5 to 20 cmH₂O and holding for 20 seconds. After recruitment, the standard ventilation group will continue with the initial ventilator settings until the end of the surgery. Patients will be ventilated in volume-controlled ventilation (VCV) mode.
  Arms: Standart Ventilation

SUMMARY:
Postoperative pulmonary complications are a frequent cause of morbidity following lumbar stabilization surgery. Conventional ventilation strategies may not adequately reflect intraoperative changes in respiratory mechanics, potentially leading to impaired postoperative pulmonary function. Dynamic compliance-guided ventilation provides a real-time, individualized approach by adjusting ventilatory parameters according to lung compliance.

This prospective randomized controlled study aims to evaluate the effects of dynamic compliance-guided ventilation compared with standard ventilation strategies on postoperative pulmonary function in patients undergoing lumbar stabilization surgery. Eligible patients will be randomly assigned to either the compliance-guided group or the conventional ventilation group.

In this study, the investigators aim to prospectively compare ventilation with the dynamic compliance (Cdyn) approach-one of the lung-protective ventilation strategies-with conventional ventilation methods in patients undergoing surgery in the prone position. The primary outcome will be evaluated using a modified lung ultrasound scoring system based on the most severely affected regions of aeration loss. Secondary objectives include the assessment of intraoperative hemodynamics, respiratory mechanics, and the effects on postoperative pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lumbar stabilization in the prone position

Exclusion Criteria:

* Patients with ASA classification IV or higher
* Patients with obesity (BMI>30) or cachexia (BMI<18)
* Allergy to standard medications used during general anesthesia
* Contraindications to PEEP (high intracranial pressure, bronchopleural fistula, hypovolemic shock, right heart failure)
* Previous lung surgery (any)
* Known serious heart disease defined as New York Heart Association class III or higher
* Patients with severe asthma and COPD
* Acute myocardial infarction within the last 12 months before surgery
* Neuromuscular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Modified Lung Ultrasound Score | baseline, postoperative 1th hour, postoperative 24th hour
  The assessment will be performed using the Modified Lung Ultrasound Scoring system. The scale ranges from a minimum of 0 to a maximum of 36 points. A score of 0 indicates normal aeration in all zones, while a score of 36 represents the worst possible aeration loss. Higher scores indicate a worse outcome (increased lung aeration loss/atelectasis).

SECONDARY OUTCOMES:
Incidence postoperative pulmonary complications(PPC) | postoperative first 7 days
  Number of participants with at least one postoperative pulmonary complication (including atelectasis, pneumonia, bronchospasm, hypoxemia, or reintubation) within the first 7 days after surgery.
  Percentage of participants
Intraoperative Dynamic Compliance (Cdyn) | intraoperative
  Mean dynamic respiratory compliance measured during the intraoperative period. Unit of Measure: mL/cmH2O
Intraoperative Plateau Pressure (Pplat) | intraoperative
  Mean airway plateau pressure measured during the intraoperative period. Unit of Measure: cmH2O
Intraoperative Driving Pressure (ΔP) | intraoperative
  Mean airway Driving Pressure measured during the intraoperative period. Unit of Measure: cmH2O
Intraoperative Peak Pressure (Ppeak) | intraoperative
  Mean airway Peak Pressure measured during the intraoperative period. Unit of Measure: cmH2O
Mean arterial pressure(MAP) | Baseline,intraoperative,1st hour postoperatively.
  Mean arterial pressure(MAP)
Heart Rate | Baseline,intraoperative,1st hour postoperatively.
  Heart Rate
Length of stay | From date of surgery until date of hospital discharge
  Hospitalization duration
Partial pressure of oxygen | Baseline, intraoperative,1st hour postoperatively.
  arterial blood oxygen partial pressure
SPO2 | Baseline,intraoperative,1st hour postoperatively.
  Measurement of non invasive oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao C, Cao H, Shen Z, Hu Y, Huang J, Shu Q, Chen Q. Comparison of volume-controlled ventilation, pressure-controlled ventilation and pressure-controlled ventilation-volume guaranteed in infants and young children in the prone position: A prospective randomized study. J Clin Anesth. 2024 Aug;95:111440. doi: 10.1016/j.jclinane.2024.111440. Epub 2024 Mar 8. PMID 38460413
- [Background] Chun EH, Baik HJ, Moon HS, Jeong K. Comparison of low and high positive end-expiratory pressure during low tidal volume ventilation in robotic gynaecological surgical patients using electrical impedance tomography: A randomised controlled trial. Eur J Anaesthesiol. 2019 Sep;36(9):641-648. doi: 10.1097/EJA.0000000000001047. PMID 31306184
- [Background] Ruszkai Z, Kiss E, Laszlo I, Bokretas GP, Vizseralek D, Vamossy I, Surany E, Buzogany I, Bajory Z, Molnar Z. Effects of intraoperative positive end-expiratory pressure optimization on respiratory mechanics and the inflammatory response: a randomized controlled trial. J Clin Monit Comput. 2021 May;35(3):469-482. doi: 10.1007/s10877-020-00519-6. Epub 2020 May 9. PMID 32388650
- [Background] Kim YJ, Kim BR, Kim HW, Jung JY, Cho HY, Seo JH, Kim WH, Kim HS, Hwangbo S, Yoon HK. Effect of driving pressure-guided positive end-expiratory pressure on postoperative pulmonary complications in patients undergoing laparoscopic or robotic surgery: a randomised controlled trial. Br J Anaesth. 2023 Nov;131(5):955-965. doi: 10.1016/j.bja.2023.08.007. Epub 2023 Sep 9. PMID 37679285